CLINICAL TRIAL: NCT05029635
Title: A Randomized, Double-blind, Placebo-controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of HMPL-523 in Treatment of Primary Immune Thrombocytopenia (ITP) in Adults(ESLIM-01 Study)
Brief Title: Phase III Study on HMPL-523 for Treatment of ITP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-523-00CH1
Record Dates: First submitted 2021-08-08; First posted 2021-08-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Primary Immune Thrombocytopenia (ITP)
Keywords: HMPL-523, sovleplenib, ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment arm (Active Comparator): Eligible subjects will be treated with planned dose of 300 mg HMPL-523 once daily for 24 weeks
  Interventions: Drug: HMPL-523
- placebo arm (Placebo Comparator): Drug: Placebo HMPL-523 matching placebo will be oral administrated once daily for 24 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HMPL-523 — HMPL-523 will be oral administrated once daily for 24 weeks
  Other Names: Sovleplenib
  Arms: treatment arm
Drug: Placebo — HMPL-523 matching placebo will be oral administrated once daily for 24 weeks .
  Arms: placebo arm

SUMMARY:
The purpose of this study is to determine whether HMPL-523 (sovleplenib) is safe and effective in the treatment of chronic Immune Thrombocytopenic Purpura (ITP).

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled phase III clinical trial in adult patients with primary immune thrombocytopenia to determine whether HMPL-523 (sovleplenib) is safe and effective in the treatment of chronic Immune Thrombocytopenic Purpura (ITP)

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of written informed consent form;
2. Male or female aged 18~75 years;
3. Performance Status score [Eastern Cooperative Oncology Group (ECOG) score] 0~1;
4. Having been diagnosed as ITP prior to randomization, and duration of disease is more than 6 months;
5. Intolerance or insufficient response, or recurrence after at least one anti-ITP standard drug therapy;
6. Patients must have a history of response to previous ITP therapy;
7. One combined anti-ITP therapy is allowed in this study, however, the following criteria need to be met:

   1. The dose of glucocorticoid has been stable for 4 weeks prior to randomization (<20 mg Prednisone equivalent);
   2. The dose of Danazol has been stable for 3 months prior to randomization;
   3. The dose of immunosuppressant (only including Azathioprine, Ciclosporin A, Mycophenolate mofetil) has been stable for 3 months prior to randomization.
8. The condition is relatively stable; WHO bleeding scale grade is 0-1; no emergency treatment is expected within 2 weeks as judged by investigators.
9. The laboratory examinations need to meet the following conditions (no treatment for this abnormal variable is given within one week prior to blood collection):

   1. Average platelet count <30×10^9 /L (and none > 35×10^9 /L unless as a result of rescue therapy) from at least 3 qualifying counts;
   2. Hemoglobin ≥100 g/L, neutrophil count >1.5×10^9/L;
   3. Total bilirubin (TBIL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤1.5×upper limit of normal (ULN);
   4. Serum creatinine concentration ≤1.5×ULN and creatinine clearance ≥50 mL/min;
   5. Serum amylase and lipase ≤1.5×ULN;
   6. International normalized ratio (INR), activated partial thromboplastin time (APTT) not exceeding 20% of normal range.
10. Male or female patients of childbearing potential must agree to use effective contraceptive methods during the study and within 90 days after last dose of study drug, e.g., double barrier contraceptive method, condom, oral or injectable contraceptives, intrauterine device, etc. Postmenopausal women (>50 years old and no menses for >1 year) and surgically sterilized women are not subject to this condition.

Exclusion Criteria:

1. Evidence on the presence of secondary causes of immune thrombocytopenia;
2. Clinically serious hemorrhage requiring immediate adjustment of platelet (e.g., hypermenorrhea with significantly decreased hemoglobin);
3. Clinically symptomatic gastrointestinal hemorrhage within 6 months prior to screening visit (e.g., haematemesis, tarry stool, however, the positive occult blood test without any sign or symptom of gastrointestinal hemorrhage will not be considered as "clinically symptomatic", or hemorrhoids hemorrhage is one exception);
4. known history of vital organ transplantation or hematopoietic stem cell / bone marrow transplantation;
5. Has received live vaccine within 8 weeks prior to Day 1 (baseline visit); or plan for immunization with live vaccine during the study;
6. Splenectomy within 12 weeks prior to randomization;
7. Major surgery within 4 weeks prior to the randomization, or plan for major elective surgery during the study;
8. Previous history of malignant tumors (except for the basal cell carcinoma of skin or cervical carcinoma in situ that have been cured);
9. History of important arterial / venous embolic disease;
10. Intracranial hemorrhage within 6 months before screening visit;
11. History of serious cardiovascular disease (e.g., grade III/IV congestive heart failure, arrhythmia or angina pectoris requiring drug therapy, unstable angina pectoris, intracoronary stent implantation, angioplasty or coronary artery bypass grafting, or QTc ≥450 ms);
12. Hypertension that can not be controlled with drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
13. Previous history of serious gastrointestinal disease, such as dysphagia, active gastric ulcer, inability to take drugs orally or absorption disorder for oral drugs;
14. Human immunodeficiency virus (HIV) infection, or hepatitis B (in case of positive HBsAg or HBcAb, positive HBV DNA needs to be determined), or hepatitis C (positive HCV RNA), or liver cirrhosis;
15. Significant active infection that is not controlled clinically (e.g., sepsis, pneumonia or abscess), or serious infection within 6 weeks prior to randomization (leading to hospitalization or requiring treatment with antibiotic injections);
16. Has received rescue therapy for ITP within 2 weeks prior to randomization; Has received the treatment for the objective of increasing platelet within 4 weeks prior to randomization (including but not limited to glucocorticoid, thrombopoietin, thrombopoietin receptor agonist, Cyclosporine A, Mycophenolate mofetil, etc.), except those meeting the inclusion criterion 7;
17. Having received Rituximab within 14 weeks prior to randomization;
18. Having received traditional Chinese medicine within 1 week prior to randomization;
19. Requiring long-term/continuous use of the drugs that may affect platelet function [including but not limited to aspirin, Clopidogrel, ticagrelor, NSAIDs, etc.], or anticoagulants;
20. Intake of potent CYP3A inhibitor or inducer, as well as sensitive or narrow therapeutic window substrates of CYP3A, CYP1A2 or CYP2B6 two weeks (three weeks for Hypericum perforatum) or 5 half-lives prior to randomization (whichever is longer);
21. Having participated in the clinical study for drugs or invasive medical device 4 weeks prior to randomization (or within 5 half-lives of the study drug prior to randomization, whichever is longer);
22. Having received spleen tyrosine kinase Syk inhibitor (e.g., Fostamatinib) previously;
23. Known allergy to the active ingredient or excipient of study drug;
24. Presence of serious psychological or mental disorder;
25. Alcoholic or drug abuser;
26. Female patients in pregnancy or breast feeding;
27. Being unsuitable to participate in this study, as considered by investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2021-10-27 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
the durable response rate in the primary study | treatment period Week14-Week24
  Platelet count ≥50×10^9 /L on at least 4 of 6 scheduled visits of Week14-Week24 in the primary study

SECONDARY OUTCOMES:
the overall response rate in the primary study | treatment period Week1-Week24 in the primary study
  At least one platelet count ≥50×10^9 /L (except that induced by the rescue therapy) in the 24-week double-blind treatment period
Incidence of treatment emergent adverse events | treatment period Week1-Week24 in the primary study
  Adverse events classified according to NCI CTCAE version 5.0
Plasma concentration at steady state 2 hours post dose (C2h,ss) | treatment period Week1-Week24 in the primary study
  Plasma concentration of HMPL-523 and its main metabolites at steady state 2 hours post dose (C2h,ss) will be determined.
Plasma concentration at steady state 2 hours post dose (C4h,ss) | treatment period Week1-Week24 in the primary study
  Plasma concentration of HMPL-523 and its main metabolites at steady state 4 hours post dose (C4h,ss) will be determined.
Plasma concentration at steady-state trough concentration (Cmin,ss) | treatment period Week1-Week24 in the primary study
  Plasma concentration of HMPL-523 and its main metabolites at steady-state trough concentration (Cmin,ss) will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Renchi Yang, professor, Principal Investigator — offices director
Locations (37):
- China (37):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated hospital of USTC, Hefei, Anhui
  - Beijing Chaoyang Hospital of Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - People's Hospital of Peking University, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Southern Hospital of Southern Medical University, Guangzhou, Guangdong
  - The Second People's Hospital Of Shenzhen, Shenzhen, Guangdong
  - The First Affiliated Hospital Of GuangXi Medical University, Nanning, Guangxi
  - The First Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Affiliated Hospital of North China University of Technology, Tangshan, Hebei
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The Affiliated Huai'an No.1 People's Hospital of Nanjing Medical University, Huai'an, Nanjing Province
  - Qinghai province people's hospital, Xining, Qinghai
  - Jinan Central Hospital Affilated to Sandong University, Jinan, Shandong
  - LiaoCheng People's Hospital, Liaocheng, Shandong
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Jinshan Hospital Affiliated To Fudan University, Shanghai, Shanghai Municipality
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - The second hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - West China Hospital，Sichuan University, Chengdu, Sichuan
  - The First Affilicated Hospital of Xinjiang Medical University, Ürümqi, The Xinjiang Uygur Autonomous Region
  - Blood Institute of the Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial Hospital of Chinese Medicine, Hangzhou, Zejiang Province

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Y, Liu X, Zhou H, Wang S, Huang R, Wang Y, Du X, Sun J, Zhou Z, Yan Z, Chen W, Wang W, Liu Q, Zeng Q, Gong Y, Yin J, Shen X, Ye B, Chen Y, Xu Y, Sun H, Cheng Y, Liu Z, Wang C, Yuan G, Zhang X, Li X, Cheng P, Guo X, Jiang Z, Yang F, Yang L, Luo C, Xiao T, Fu S, Yin H, Guo X, Xu Q, Fan S, Shi MM, Su W, Mei H, Yang R. Efficacy and safety of sovleplenib (HMPL-523) in adult patients with chronic primary immune thrombocytopenia in China (ESLIM-01): a randomised, double-blind, placebo-controlled, phase 3 study. Lancet Haematol. 2024 Aug;11(8):e567-e579. doi: 10.1016/S2352-3026(24)00139-X. Epub 2024 Jun 14. PMID 38885672